CLINICAL TRIAL: NCT04926311
Title: Efficiency of Speech and Language Intervention on Achievement of Children With Developmental Language Disorder
Acronym: DYSPHADEV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0052
Record Dates: First submitted 2021-06-08; First posted 2021-06-15 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Language Development Disorders; Speech and Language Disorder; Therapy
Keywords: Language Development Disorders; Speech and Language Disorder; Academic outcomes
MeSH Terms: conditions — Language Development Disorders; Speech; Language Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Developmental Language Disorder patients

SUMMARY:
Children with Developmental Language Disorder (DLD) have many linguistic difficulties in syntax, lexicon, morphology and phonology. Frequently, they also present co-occurrent (or comorbidities) impairments which further impaired school learning. Thus, they have poor academic outcomes and many of these children have been maintained at least one time in a classroom, sometime more.

The purpose of this project is to determine which modalities of speech and language therapy are the more efficient on academic outcomes of children with DLD. The main modalities that will be studied are the duration of speech and language intervention, the age at which begins the intervention and the intensity (number of intervention sessions per week).

ELIGIBILITY:
Inclusion Criteria:

* patients Have been diagnosed in the University Hospital of Amiens-Picardie with a Developmental Language Disorder
* patients must be aged 12 or older,
* patients must be agreed answering the questionnaire

Exclusion Criteria:

* Children with a neurological pathology or handicap as epilepsy, cerebral palsy, sequelae of severe brain injury (traumatic or ischemic or inflammatory...)
* patients with a severe mental retardation
* patients with autism
* patients with bipolar illness
* patients with psychosis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients agreed to participate in the study will respond by phone to a questionnaire providing information on modalities of speech and langage intervention therapy, their course of school and academic studies, potentially associated developmental disorders and their management. Analysis will focused on the effects of speech and langage therapy modalities (intensity, age onset, duration), comorbidities and their management if concerned, special education resource teacher or specialized board-level support during the school trajectory on the school grade repetition in the patients of the study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Number of repeated school year according length of language therapy (number of days) | one day
  Number of repeated school year according length of language therapy

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No